CLINICAL TRIAL: NCT06398561
Title: Peer-led Intervention for Individuals With Major Depression.
Acronym: SUPEERmood
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GH2023/07
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Depressive Disorder, Major
Keywords: peer-leader; promotion; mental health; depression; peer to peer; health education
MeSH Terms: conditions — Depressive Disorder, Major; Psychological Well-Being; Depression; Health Education

STUDY DESIGN:
Intervention Model Description: A two-branch randomized clinical trial will be carried out, in which one branch will receive the intervention based on a peer support program (Active Patient Program) and the other branch will receive information and exercises aimed at improving their mental health through a validated App, free and in its Spanish version, called "COGITO", which consists of planning exercises based on cognitive-behavioral therapy. The App to be used can be found for free by accessing the following link: https://apps.apple.com/us/app/cogito-mct/id1557322291 (for Apple devices) https://play.google.com/store/apps/details?id=de.uke.cogitoapp&hl=en_US&pli=1 (for Android devices).
  A measurement of the study variables will be carried out through validated instruments at the beginning of the program, another one at the end of the six sessions (6 weeks), 6 and 12 months after the last session.
Who Masked: Outcomes Assessor
Masking Description: We randomized the participants across the informatic program named RedCap. Only was masking the outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Active Patient Program intervention (Experimental): The intervention consists of carrying out the six sessions of the Active Patient Program by peers. The sessions have a duration of 2 hours/week during 6 weeks. It is aimed at patients with a diagnosis of major depression and they will undergo 4 evaluations, one before, one at the end of the sessions and two more at 6 and 12 months after the end of the sessions.
  Interventions: Behavioral: Active Patient Program
- Control: Use App COGITO (Active Comparator): the control consists of the regular use (30 minutes daily) of the COGITO App that will guide the participant in the performance of exercises to improve depressive symptomatology. The time of use is equivalent to the time invested in the sessions.
  The same evaluations will be carried out as in the experimental group (previous evaluation, at the end of the sessions (6 weeks) and two more at 6 and 12 months after the end of the sessions.
  Interventions: Behavioral: Active Patient Program

INTERVENTIONS:
Behavioral: Active Patient Program — The Active Patient Program is a peer-leader intervention that consist of training patients with a chronic disease or mental health illness for improve the symptoms of that pathology.
  Training is carried out in groups of about 12-15 patients and usually has 2 patient trainers. These patients lead the sessions through the theoretical content they have integrated, motivation, group leadership, exchange of experiences and promotion of communication. In this way they favor problem-solving by the patients who attend the sessions, thus improving their self-management and self-efficacy.
  In the group formed by patients who are trainers and patients who benefit from the sessions, a climate of trust is created that favors the expression of emotions on both sides, empathy and assertiveness. In addition to fostering socio-affective bonds between the participants and increasing perceived social and emotional support.

SUMMARY:
Objective: To evaluate the efficacy of an adjuvant intervention based on a peer support program in the reduction of depressive symptomatology versus an online intervention in people with major depression in Primary Care Mental Health Units in Mallorca.

Design: Randomized clinical trial of two branches in a Mental Health Unit of Mallorca, where one branch will receive an adjuvant intervention based on a peer support program (Active Patient Program) and another branch (control) will receive information and exercises aimed at improving their mental health through the COGITO App, designed and validated for this purpose.

Scope and study subjects: The scope of the study will be the consultations of the Mental Health Unit (MHU) of Primary Care in Mallorca. The study subjects will be patients of these units who meet the criteria for Major Depression. The mental health professionals of the MHU will be in charge of recruiting participants who meet the inclusion and exclusion criteria. The required sample will be 70 subjects, 35 in each branch.

Variables: The main dependent variable is depressive symptomatology, measured through the Beck Depression Inventory (BDI-II). As secondary variables, quality of life and adherence to treatment will be included.

Data analysis: All analyses will be carried out using the SPSS statistical program. An intention-to-treat (ITT) analysis will be performed. The efficacy of the intervention (reduction of depressive symptoms (BDI-II)) will be assessed by a general linear model (ANOVA) at 6 weeks, 6 and 12 months, adjusted for baseline values.

DETAILED DESCRIPTION:
Material and methods Type of study A two-branch randomized clinical trial will be conducted, in which one branch will receive the intervention based on a peer support program (Active Patient Program) and another branch will receive information and exercises aimed at improving their mental health through a validated App, free and in its Spanish version, called "COGITO", which consists of planning exercises based on cognitive-behavioral therapy. The App to be used can be found for free by accessing the following link: https://apps.apple.com/us/app/cogito-mct/id1557322291 (for Apple devices) https://play.google.com/store/apps/details?id=de.uke.cogitoapp&hl=en_US&pli=1 (for Android devices).

Scope of the study The consultations of the Mental Health Unit (MHU) will be the site from which the subjects will be recruited. The MHU are outpatient and community facilities of the mental health network of the Balearic Islands, where people with mental health problems are followed up. They consist of a multidisciplinary team of psychiatry, psychology, mental health nursing and social work professionals. In addition to the administrative staff of these units.

Definition of study subjects The study subjects will be those persons suffering from Major Depressive Disorder and who are currently under follow-up with one of the professionals of the MHU.

Recruitment of participants Recruitment will be done through the medical records of each nurse, psychiatrist, psychologist or social worker of the USM with current follow-up and/or active diagnostic label of Major Depressive Disorder (according to ICD or DSM criteria) in the Primary Care Information System (e-SIAP).

An initial interview will be carried out by the research staff in collaboration with the health care staff of the reference MHU to verify compliance with the inclusion criteria for the study.

Justification of sample size Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 35 subjects in the intervention group (Active Patient) and 35 in the control group are required to detect a difference equal to or greater than 6 units in the Beck Depression Inventory (BDI-II). The common standard deviation is assumed to be 8. A loss-to-follow-up rate of 20% has been estimated (Castro LS et al. Psychiatry Res. 2013;210(3):906-12). Therefore, a total of 70 participants will be needed.

Primary and secondary variables. The primary dependent variable is depressive symptomatology measured by validated BDI-II.

The secondary dependent variables are quality of life and adherence to prescribed treatment. The main independent variable is the assigned group.

Other independent or control variables taken into account in this study are sociodemographic variables (age, gender, marital status, diagnostic label, year of diagnosis, educational level, pharmacological treatment, psychotherapy treatment, USM of reference, profession, comorbidities, current employment situation).

Description of the intervention

1. Recruitment and training of active patient trainers:

   Recruitment will be carried out by MHU professionals, through any device of the mental health network or through patients' associations and/or citizens' associations.

   The trainer patients must meet the following requirements according to the current protocol of the Active Patient Program, evaluated through the interview, the scales and questionnaires that the program stipulates in its action guide. All the information regarding this aspect can be found in detail at the following link: https://docusalut.com/handle/20.500.13003/18170.
2. Recruitment of participants The recruitment of the study subjects will be carried out by the multidisciplinary team of the MHU (psychiatrists, psychologists, nurses and/or social workers of each center). Once the sample has been recruited, an initial interview will be conducted by the staff of the Active Patient Program team to explain the procedure and assess whether the selected persons accept their participation and meet the inclusion criteria described above.
3. Randomization Once the necessary sample has been obtained, the participants will be randomized in a 1:1 ratio.Pseudo-anonymity of the data is guaranteed, since each participant will be identified with a numerical code that will not include any personal data.
4. Development of the intervention- Intervention group for patients benefiting from the Active Patient Program training.

   The training will consist of a workshop of 6 sessions of 2 hours each, following the model described in the protocol of the Active Patient Program but adapted to Major Depressive Disorder.

   The adaptation of this guide will be carried out by a group of professionals, from different disciplines, experts in mental health. Once the guide has been produced, it will be sent to people of reference in the field of depressive disorders at a national level, so that they can proceed to its revision.

   The sessions that will guide us in the preparation of the Major Depressive Disorder workshop are detailed in Annex I.- Control group through the COGITO App.The control group will receive a guideline of exercises guided through the COGITO App based on cognitive-behavioral therapy (CBT). The duration of the use of this App will be the same as the intervention of the Active Patient program (6 weeks), having to comply with a pattern of use of the App of 20 minutes daily in order to match the time dedicated to the intervention. Thanks to the design of the App, its use can be counted through the history of the exercises, as well as the appearance of warnings when the use is low.Daily reminders can also be activated to incentivize it.
5. Evaluation:

A pre-intervention evaluation will be carried out at the beginning of the intervention in both groups, another one at the end of the program sessions (6 weeks) and two post- evaluations at 6 and 12 months after completion.

The degree of depressive symptomatology, the quality of life and the degree of adherence to the prescribed treatment will be measured by means of valid instruments.

ELIGIBILITY:
Selection and withdrawal of subjects

Inclusion criteria:

* People over 18 years of age.
* Attending consultations with any of the professionals in the USM mental health network.
* Having an active diagnostic label of Major Depressive Disorder, according to ICD or DSM criteria in the Primary Care e-SIAP program or meeting MINI TRAS criteria after individual interview for Major Depressive Episode.

Exclusion criteria

* People who present mental health disorders associated with a depressive disorder and who are in the acute phase of the disease.
* People who are not under active follow-up with any of the professionals of the USM.
* People with mobility problems and / or displacement to the health center.
* People suffering from another disease affecting the CNS (organic brain pathology or who have suffered a severe head injury, onset dementia or any other neurodegenerative disease, etc.).
* People with presence of uncontrolled serious medical, infectious or degenerative disease, which may interfere with affective symptomatology.
* People with significant risk of suicide according to medical criteria, assessed through follow-up interviews conducted by mental health professionals of reference.
* People with any medical, psychological and/or social problem that could seriously interfere with the patient's participation in the study.
* People who are legally incapacitated to make health decisions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of an adjuvant intervention based on a peer-leader program (Active Patient Program) | 12 months
  To measure the efficacy of an adjuvant intervention based on a peer-leader program (Active Patient Program) for the reduction on 6 points the depressive sympthoms with the Beck Depression Inventory in a sample of 70 people with Major Depression versus an online intervention in Primary Care Mental Health Units in Mallorca.Using Beck Depression Inventory (BDI-II) we want to know if the intervention can reduce the depressive symptoms.

SECONDARY OUTCOMES:
To analyze the efficacy of the proposed intervention on adherence to the prescribed treatment of people with Major Depression. | 12 months
  To measure the adherence to psychiatric treatment, we use the Drug Attitude Inventory (DAI-10) questionnaire. In a sample of 70 people with Major Depression, we want to know if the intervention can improve the treatment adherence of life of the participants.
To evaluate the effect of intervention on the quality of life of people with Major Depression. | 12 months
  To analyze the life-quality, we use the EuroQoL-5D questionnaire and measure the differences in the baseline life-quality and the following visits post intervention and post control in a sample of 70 people with Major Depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Xandra González García, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] World Health Organization. Depression 2021. Available from: https://www.who.int/es/news-room/fact-sheets/detail/depression.
- [Result] Global Health Data Exchange. Global Health Data Exchange (GHDx) 2021. Available from:http://ghdx.healthdata.org/gbd-results-tool?params=gbd-api-2019-permalink/442c335139ab11cec605591fd4141f0d.
- [Result] Zhang Z, Jackson SL, Gillespie C, Merritt R, Yang Q. Depressive Symptoms and Mortality Among US Adults. JAMA Netw Open. 2023 Oct 2;6(10):e2337011. doi: 10.1001/jamanetworkopen.2023.37011. PMID 37812418
- [Result] Garcia A, Yanez AM, Bennasar-Veny M, Navarro C, Salva J, Ibarra O, Gomez-Juanes R, Serrano-Ripoll MJ, Olivan B, Gili M, Roca M, Riera-Serra P, Aguilar-Latorre A, Montero-Marin J, Garcia-Toro M. Efficacy of an adjuvant non-face-to-face multimodal lifestyle modification program for patients with treatment-resistant major depression: A randomized controlled trial. Psychiatry Res. 2023 Jan;319:114975. doi: 10.1016/j.psychres.2022.114975. Epub 2022 Nov 22. PMID 36442318
- [Result] Grupo de trabajo de la Guía de Práctica Clínica sobre el Manejo de la Depresión en el Adulto. Guía de Práctica Clínica sobre el Manejo de la Depresión en el Adulto.: Ministerio de Sanidad, servicios Sociales e Igualdad. Agencia de Evaluación de Tecnnologías Sanitarias de Galicia (avalia-t); 2014.
- [Result] Salehi I, Hosseini SM, Haghighi M, Jahangard L, Bajoghli H, Gerber M, Puhse U, Holsboer-Trachsler E, Brand S. Electroconvulsive therapy (ECT) and aerobic exercise training (AET) increased plasma BDNF and ameliorated depressive symptoms in patients suffering from major depressive disorder. J Psychiatr Res. 2016 May;76:1-8. doi: 10.1016/j.jpsychires.2016.01.012. Epub 2016 Jan 25. PMID 26859236
- [Result] Wong VW, Ho FY, Shi NK, Sarris J, Chung KF, Yeung WF. Lifestyle medicine for depression: A meta-analysis of randomized controlled trials. J Affect Disord. 2021 Apr 1;284:203-216. doi: 10.1016/j.jad.2021.02.012. Epub 2021 Feb 5. PMID 33609955
- [Result] Eiroa-Orosa FJ, Sanchez-Moscona C. Implementing the figure of peer support workers in mental health: an international perspective from the context of its implementation in Catalonia. Salud Colect. 2023 Jan 23;19:e4252. doi: 10.18294/sc.2023.4252. English, Spanish. PMID 37311138
- [Result] Davidson L, Bellamy C, Guy K, Miller R. Peer support among persons with severe mental illnesses: a review of evidence and experience. World Psychiatry. 2012 Jun;11(2):123-8. doi: 10.1016/j.wpsyc.2012.05.009. PMID 22654945
- [Result] Smit D, Miguel C, Vrijsen JN, Groeneweg B, Spijker J, Cuijpers P. The effectiveness of peer support for individuals with mental illness: systematic review and meta-analysis. Psychol Med. 2023 Aug;53(11):5332-5341. doi: 10.1017/S0033291722002422. Epub 2022 Sep 6. PMID 36066104
- [Result] Naslund JA, Aschbrenner KA, Marsch LA, Bartels SJ. The future of mental health care: peer-to-peer support and social media. Epidemiol Psychiatr Sci. 2016 Apr;25(2):113-22. doi: 10.1017/S2045796015001067. Epub 2016 Jan 8. PMID 26744309
- [Result] Sastre Perea MJ, Vidal Thomàs MC, Cáceres Teijeiro Y, Moreno Sancho ML, Miguelez Chamorro A, Font Oliver MA, et al. Programa Pacient Actiu de les Illes Balears. Palma: Servei de Salut de les Illes Balears; 2018.
- [Result] Peer Support Canada. Guiding connection Strategic Plan 2022-2027. Canada; 2022. Available from: https://peersupportcanada.ca/wp-content/uploads/2022/11/Peer-Support-Canada-Strategic-Plan-1.pdf
- [Result] Cherrington AL, Khodneva Y, Richman JS, Andreae SJ, Gamboa C, Safford MM. Impact of Peer Support on Acute Care Visits and Hospitalizations for Individuals With Diabetes and Depressive Symptoms: A Cluster-Randomized Controlled Trial. Diabetes Care. 2018 Dec;41(12):2463-2470. doi: 10.2337/dc18-0550. Epub 2018 Oct 29. PMID 30373734
- [Result] Prevatt BS, Lowder EM, Desmarais SL. Peer-support intervention for postpartum depression: Participant satisfaction and program effectiveness. Midwifery. 2018 Sep;64:38-47. doi: 10.1016/j.midw.2018.05.009. Epub 2018 May 31. PMID 29908406
- [Result] Liu T, Leung DKY, Lu S, Kwok WW, Sze LCY, Tse SSK, Ng SM, Wong PWC, Lou VWQ, Tang JYM, Wong DFK, Chan WC, Kwok RYK, Lum TYS, Wong GHY. Collaborative community mental health and aged care services with peer support to prevent late-life depression: study protocol for a non-randomised controlled trial. Trials. 2022 Apr 11;23(1):280. doi: 10.1186/s13063-022-06122-1. PMID 35410292
- [Result] Simmons MB, Cartner S, MacDonald R, Whitson S, Bailey A, Brown E. The effectiveness of peer support from a person with lived experience of mental health challenges for young people with anxiety and depression: a systematic review. BMC Psychiatry. 2023 Mar 24;23(1):194. doi: 10.1186/s12888-023-04578-2. PMID 36964523
- [Result] Byrom N. An evaluation of a peer support intervention for student mental health. J Ment Health. 2018 Jun;27(3):240-246. doi: 10.1080/09638237.2018.1437605. Epub 2018 Feb 16. PMID 29451411
- [Result] Mahlke CI, Priebe S, Heumann K, Daubmann A, Wegscheider K, Bock T. Effectiveness of one-to-one peer support for patients with severe mental illness - a randomised controlled trial. Eur Psychiatry. 2017 May;42:103-110. doi: 10.1016/j.eurpsy.2016.12.007. Epub 2016 Dec 28. PMID 28364685
- [Result] Lauridsen S, Nielsen MBD, Kusier AO, Cloos CO, Jensen MP, Andersen S, Thygesen LC, Folker AP. Implementing a peer-to-peer, self-management intervention for young people with depression and anxiety in Denmark. BMC Psychol. 2022 Mar 16;10(1):70. doi: 10.1186/s40359-022-00777-w. PMID 35296363
- [Result] Richard J, Rebinsky R, Suresh R, Kubic S, Carter A, Cunningham JEA, Ker A, Williams K, Sorin M. Scoping review to evaluate the effects of peer support on the mental health of young adults. BMJ Open. 2022 Aug 4;12(8):e061336. doi: 10.1136/bmjopen-2022-061336. PMID 35926986
- [Result] Thomas EC, Simmons MB, Mathai C, Salzer MS. Peer-Facilitated Decision Making in Mental Health: Promises, Pitfalls, and Recommendations for Research and Practice. Psychiatr Serv. 2023 Apr 1;74(4):401-406. doi: 10.1176/appi.ps.20220086. Epub 2022 Sep 27. PMID 36164774
- [Result] Valenstein M, Pfeiffer PN, Brandfon S, Walters H, Ganoczy D, Kim HM, Cohen JL, Benn-Burton W, Carroll E, Henry J, Garcia E, Risk B, Kales HC, Piette JD, Heisler M. Augmenting Ongoing Depression Care With a Mutual Peer Support Intervention Versus Self-Help Materials Alone: A Randomized Trial. Psychiatr Serv. 2016 Feb;67(2):236-9. doi: 10.1176/appi.ps.201400454. Epub 2015 Sep 15. PMID 26369884
- [Result] Mantani A, Kato T, Furukawa TA, Horikoshi M, Imai H, Hiroe T, Chino B, Funayama T, Yonemoto N, Zhou Q, Kawanishi N. Smartphone Cognitive Behavioral Therapy as an Adjunct to Pharmacotherapy for Refractory Depression: Randomized Controlled Trial. J Med Internet Res. 2017 Nov 3;19(11):e373. doi: 10.2196/jmir.8602. PMID 29101095
- [Derived] Gonzalez-Garcia X, Moreno-Sancho ML, Roa-Diez P, Caceres-Tejeiro Y, Flowers SA, de Montes CG, Bennasar-Veny M, Garcia-Toro M, Yanez AM. Peer-led intervention for individuals with major depression: study protocol for a randomized controlled trial (SUPEERMood). BMC Psychiatry. 2024 Sep 30;24(1):639. doi: 10.1186/s12888-024-06094-3. PMID 39350120